CLINICAL TRIAL: NCT04571619
Title: A Randomized Clinical Trial to Evaluate Non-Pharmacologic and Pharmacologic Approaches for Reducing Pain and Opioid Use Among Patients Treated With Maintenance Hemodialysis
Brief Title: HOPE Consortium Trial to Reduce Pain and Opioid Use in Hemodialysis
Acronym: HOPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Hennepin Health Care (Unknown); New York University (Other); Massachusetts General Hospital (Other); University of Illinois at Chicago (Other); University of Pittsburgh (Other); University of Washington (Other); University of New Mexico (Other); Rogosin Institute (Unknown); Vanderbilt University Medical Center (Other); West Virginia University (Other); Yale University (Other); Durham VA Health Care System (U.S. Federal Agency); VA Portland Healthcare System (Unknown); West Haven VA Medical Center (Unknown); University of Pennsylvania (Other); Dallas VA Medical Center (U.S. Federal Agency); VA New York Harbor Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HOPE; U01DK123813 (NIH); U01DK123786 (NIH); U01DK123787 (NIH); U01DK123812 (NIH); U01DK123814 (NIH); U01DK123816 (NIH); U01DK123817 (NIH); U01DK123818 (NIH); U01DK123821 (NIH)
Record Dates: First submitted 2020-09-15; First posted 2020-10-01 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-06

CONDITIONS: End Stage Renal Disease; Chronic Pain; Opioid Dependence
Keywords: hemodialysis; pain; opioids; pain coping skills
MeSH Terms: conditions — Kidney Failure, Chronic; Chronic Pain; Opioid-Related Disorders; Pain | interventions — Buprenorphine

STUDY DESIGN:
Intervention Model Description: Sequential multiple assignment design with a randomized component followed by a non-randomized component
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain Coping Skills Training (Active Comparator): The PCST intervention will focus primarily on reducing pain interference in daily activities and improving pain self-management skills. For participants with recent or current opioid use, the PCST intervention will include motivational interviewing aimed at reducing opioid use. During Weeks 1 - 12 the PCST will be delivered by coaches via telehealth (video). During Weeks 13 - 24, the Interactive Voice Response (IVR) will be delivered via telephone. The telehealth component will consist of weekly sessions, each lasting 45-50 minutes. The IVR content, intended to enhance and sustain the effects of the coach-led session, will be delivered with daily telephone interactions, each lasting approximately 5 minutes. Both components of the intervention will be available in English and Spanish.
  Interventions: Behavioral: Pain Coping Skills Training (PCST); Drug: Buprenorphine
- Usual Care (Other): Participants in the Usual Care arm will be provided with written educational material about chronic pain and opioid medications, and available resources for treatment.
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Behavioral: Pain Coping Skills Training (PCST) — The PCST intervention will focus primarily on reducing pain interference in daily activities and improving pain self-management skills. For participants with recent or current opioid use, the PCST intervention will include motivational interviewing aimed at reducing opioid use. During Weeks 1 - 12 the PCST will be delivered by coaches via telehealth (video). During Weeks 13 - 24, the Interactive Voice Response (IVR) will be delivered via telephone. The telehealth component will consist of weekly sessions, each lasting 45-50 minutes. The IVR content, intended to enhance and sustain the effects of the coach-led session, will be delivered with daily telephone interactions, each lasting approximately 5 minutes. Both components of the intervention will be available in English and Spanish.
  Arms: Pain Coping Skills Training
Drug: Buprenorphine — At Week 24, participants who meet the eligibility criteria for the buprenorphine intervention will be encouraged to switch from their current full agonist opioid medication to the partial opioid agonist, buprenorphine. Participants who switch to Buprenorphine will be provided with individualized buprenorphine treatment recommendations. Individualized buprenorphine treatment recommendations will be made by the study buprenorphine physician based on current opioid use and other relevant factors. Participants who do not meet the Phase 2 eligibility criteria will not be offered buprenorphine. All participants will continue to be followed from Week 24 until Week 36 for ascertainment of pain, opioid use, and other outcomes to address durability of the effects of PCST, and, for those who switch to buprenorphine, to assess buprenorphine acceptability, tolerability, and efficacy as exploratory outcomes.

SUMMARY:
HOPE is a randomized clinical trial that will evaluate approaches to reducing pain and opioid use among patients with chronic pain who are receiving maintenance hemodialysis for end-stage renal disease. The hypothesis is that pain coping skills training will be effective at reducing pain and opioid use, and that buprenorphine will be acceptable and tolerable as an approach to managing physical dependence on opioids in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Undergoing in-center maintenance hemodialysis for ≥90 days
3. English- or Spanish-speaking
4. Chronic pain defined as a response of "Most days" or "Every day" to the following question: "In the past 3 months, how often have you had pain?" Answer options: Never, Some days, Most days, Every day
5. Current Pain, Enjoyment of Life and General Activity Scale (PEG) score ≥ 4
6. Willing to provide informed consent
7. Willing to allow research team to obtain opioid pharmacy refill data
8. Willing to allow research team to contact and work with their opioid prescriber

Exclusion Criteria:

1. Current opioid use disorder
2. Current use of heroin
3. Current non-opioid substance use disorder with the exception of tobacco use disorder
4. Current use of methadone, buprenorphine, or naltrexone for opioid use disorder
5. Current receipt of hospice care
6. Cognitive impairment that, in the judgement of the research team, precludes trial participation
7. Active suicidal intent
8. Unstable bipolar disorder, schizophrenia, post-traumatic stress disorder, or other psychotic disorder
9. Life expectancy < 6 months
10. Expected to receive a kidney transplant, transfer to another dialysis facility, or transition to home dialysis within 6 months
11. Current incarceration
12. Any other condition that the investigator considers precludes participation in the clinical trial

Subgroup with Current or Recent Opioid Use During eligibility screening all potential participants will have opioid use ascertained using the timeline follow back approach. The trial will enroll at least 300 participants (among the 640 total study participants) with current or recent opioid use defined as patient-reported prescription opioid use during at least 3 of the past 6 months. The number of participants in the opioid use subgroup will be monitored throughout the trial enrollment period. If the rate of enrollment into the opioid use subgroup is lower than targeted, trial enrollment will be restricted to individuals meeting the opioid use criteria as long as necessary to ensure that the total enrollment target for the trial is not met without reaching the opioid use subgroup target.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dember, MD, Principal Investigator — University of Pennsylvania
Locations (16):
- United States (16):
  - West Haven VA Healthcare System, West Haven, Connecticut
  - University of Illinois at Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of New Mexico, Albuquerque, New Mexico
  - New York University, New York, New York
  - VA NY Harbor Healthcare System, New York, New York
  - Rogosin Institute, New York, New York
  - Durham VA Healthcare System, Durham, North Carolina
  - VA Portland Healthcare System, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data will be transferred to the National Institute of Diabetes and Digestive and Kidney Diseases NIDDK) Central Repository after the trial has been completed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Dember LM, Hsu JY, Mehrotra R, Cavanaugh KL, Kalim S, Charytan DM, Fischer MJ, Jhamb M, Johansen KL, Becker WC, Pellegrino B, Eneanya ND, Schrauben SJ, Pun PH, Unruh ML, Morasco BJ, Mehta M, Miyawaki N, Penfield J, Bernardo L, Brintz CE, Cheatle MD, Doorenbos AZ, Heapy AA, Keefe FJ, Krebs EE, Kuzla N, Nigwekar SU, Schmidt RJ, Steel JL, Wetmore JB, White DM, Kimmel PL, Cukor D; HOPE Consortium. Pain Coping Skills Training for Patients Receiving Hemodialysis: The HOPE Consortium Randomized Clinical Trial. JAMA Intern Med. 2025 Feb 1;185(2):197-207. doi: 10.1001/jamainternmed.2024.7140. PMID 39786400
- [Derived] Steel JL, Brintz CE, Heapy AA, Keefe F, Cheatle MD, Jhamb M, McNeil DW, Shallcross AJ, Kimmel PL, Dember LM, White DM, Williams J, Cukor D. Adapting a pain coping skills training intervention for people with chronic pain receiving maintenance hemodialysis for end stage Kidney disease. J Behav Med. 2025 Apr;48(2):298-307. doi: 10.1007/s10865-024-00534-x. Epub 2024 Dec 3. PMID 39627496
- [Derived] Dember LM, Hsu JY, Bernardo L, Cavanaugh KL, Charytan DM, Crowley ST, Cukor D, Doorenbos AZ, Edwards DA, Esserman D, Fischer MJ, Jhamb M, Joffe S, Johansen KL, Kalim S, Keefe FJ, Kimmel PL, Krebs EE, Kuzla N, Mehrotra R, Mishra P, Pellegrino B, Steel JL, Unruh ML, White DM, Yabes JG, Becker WC; HOPE Consortium. The design and baseline characteristics for the HOPE Consortium Trial to reduce pain and opioid use in hemodialysis. Contemp Clin Trials. 2024 Jan;136:107409. doi: 10.1016/j.cct.2023.107409. Epub 2023 Dec 10. PMID 38086444

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 643 participants were randomized across 16 recruitment sites.
Pre-assignment Details: The original enrollment target was 640 participants. Permission to over-enroll was granted by the single IRB of record due to the nature of 16 recruitment sites enrolling simultaneously. The study teams did not want to have to exclude participants who had been consented and were in the screening process when the original target of 640 was reached. Therefore, 3 extra participants were enrolled as they had already been consented when the 640th participant was randomized.
Groups:
- Pain Coping Skills Training (PCST): PCST: Participants in the PCST arm will be provided with written educational material about chronic pain and opioid medications, and available resources for treatment. The PCST intervention aims to reduce pain interference and improve self-management skills. During Weeks 1-12 the PCST will be delivered by coaches via weekly video- or tele-conferencing sessions. During Weeks 13-24, Interactive Voice Response (IVR) will be delivered via daily telephone interactions, each lasting approximately 5 minutes. The IVR content is intended to enhance and sustain the effects of the coach-led session. Both components of the intervention will be available in English and Spanish.
  Buprenorphine: At Week 24, participants who meet the eligibility criteria for the buprenorphine intervention will be encouraged to switch from their full agonist opioid medication to the partial opioid agonist, buprenorphine. Participants who switch will be provided with individualized buprenorphine treatment recommendations made by a study physician based on current opioid use and other relevant factors. Participants who do not meet the Phase 2 eligibility criteria will not be offered buprenorphine. All participants will continue to be followed from Week 24 until Week 36 for ascertainment of pain, opioid use, and other outcomes to address durability of the effects of PCST, and, for those who switch to buprenorphine, to assess buprenorphine acceptability, tolerability, and efficacy as exploratory outcomes.
- Usual Care: Usual Care: Participants in the Usual Care arm will be provided with written educational material about chronic pain and opioid medications, and available resources for treatment.
  Buprenorphine: At Week 24, participants who meet the eligibility criteria for the buprenorphine intervention will be encouraged to switch from their current full agonist opioid medication to the partial opioid agonist, buprenorphine. Participants who switch to Buprenorphine will be provided with individualized buprenorphine treatment recommendations. Individualized buprenorphine treatment recommendations will be made by the study buprenorphine physician based on current opioid use and other relevant factors. Participants who do not meet the Phase 2 eligibility criteria will not be offered buprenorphine. All participants will continue to be followed from Week 24 until Week 36 for ascertainment of pain, opioid use, and other outcomes to address durability of the effects of PCST, and, for those who switch to buprenorphine, to assess buprenorphine acceptability, tolerability, and efficacy as exploratory outcomes.
Period: Phase 1
Arm/Group | Pain Coping Skills Training (PCST) | Usual Care
Started | 319 | 324
Completed | 290 | 304
Not Completed | 29 | 20
Not completed — Death | 22 | 18
Not completed — Withdrawal by Subject | 7 | 2
Period: Phase 2
Arm/Group | Pain Coping Skills Training (PCST) | Usual Care
Started | 290 | 304
Completed | 271 | 284
Not Completed | 19 | 20
Not completed — Death | 13 | 16
Not completed — Withdrawal by Subject | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Usual Care: Participants in the Usual Care arm will be provided with written educational material about chronic pain and opioid medications, and available resources for treatment.
- Total: Total of all reporting groups
Arm/Group | Pain Coping Skills Training | Usual Care | Total
Number analyzed (Participants) | 319 | 324 | 643
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 193 | 194 | 387
  >=65 years | 126 | 130 | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (12.6) | 60.4 (12.5) | 60.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 138 | 293
  Male | 164 | 186 | 350
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62 | 57 | 119
  Not Hispanic or Latino | 256 | 261 | 517
  Unknown or Not Reported | 1 | 6 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 12 | 22
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 4 | 6
  Black or African American | 160 | 148 | 308
  White | 99 | 111 | 210
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 39 | 41 | 80
Region of Enrollment [Number; unit: participants]
  United States | 319 | 324 | 643

OUTCOME MEASURES:

1. Primary Outcome: Pain Interference
Description: Pain interference as measured by the Brief Pain Index (BPI) Interference Scale. This is typically scored as the mean of the seven items. Lowest score - 0; Highest score - 10. A higher score is worse.
Time Frame: The primary outcome of pain interference will be ascertained at Week 12 coinciding with the end of the PCST weekly coaching sessions.
Population: Participants withdrew at various points during the trial. Some participants were not able to complete the PRO assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pain Coping Skills Training: PCST: Participants in the PCST arm will be provided with written educational material about chronic pain and opioid medications, and available resources for treatment. The PCST intervention aims to reduce pain interference and improve self-management skills. During Weeks 1-12 the PCST will be delivered by coaches via weekly video- or tele-conferencing sessions. During Weeks 13-24, Interactive Voice Response (IVR) will be delivered via daily telephone interactions, each lasting approximately 5 minutes. The IVR content is intended to enhance and sustain the effects of the coach-led session. Both components of the intervention will be available in English and Spanish.
  Buprenorphine: At Week 24, participants who meet the eligibility criteria for the buprenorphine intervention will be encouraged to switch from their full agonist opioid medication to the partial opioid agonist, buprenorphine. Participants who switch will be provided with individualized buprenorphine treatment recommendations made by a study physician based on current opioid use and other relevant factors. Participants who do not meet the Phase 2 eligibility criteria will not be offered buprenorphine. All participants will continue to be followed from Week 24 until Week 36 for ascertainment of pain, opioid use, and other outcomes to address durability of the effects of PCST, and, for those who switch to buprenorphine, to assess buprenorphine acceptability, tolerability, and efficacy as exploratory outcomes.
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 318 | 324
score on a scale
  Baseline | 6.26 (2.02) | 6.45 (2.13)
  Week 12 | 5.09 (2.37) | 5.75 (2.55)

2. Secondary Outcome: Pain Intensity
Description: Pain intensity as measured by the Brief Pain Index (BPI) Severity Scale. Lowest score - 0; Highest score - 40. A higher score is worse.
Time Frame: Weeks 12, 24, and 36
Population: Participants withdrew at various points during the study. Some participants were not able to complete the PRO assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
score on a scale
  Baseline: number analyzed (Participants) | 318 | 322
  Baseline | 5.83 (2.05) | 5.98 (2.13)
  Week 12: number analyzed (Participants) | 282 | 290
  Week 12 | 4.95 (2.32) | 5.38 (2.24)
  Week 24: number analyzed (Participants) | 258 | 263
  Week 24 | 4.64 (2.44) | 5.21 (2.31)
  Week 36: number analyzed (Participants) | 248 | 254
  Week 36 | 4.74 (2.49) | 5.10 (2.46)

3. Secondary Outcome: Pain Catastrophizing
Description: Pain catastrophizing will be measured using the Pain Catastrophizing Scale (PCS) Short Form (SF) 6. Lowest score - 0; Highest score - 24. A higher score is worse.
Time Frame: Weeks 12, 24, and 36
Population: Participants withdrew at various points throughout the study, and some participants were unable to complete the PRO assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
score on a scale
  Baseline: number analyzed (Participants) | 316 | 319
  Baseline | 15.5 (5.61) | 15.5 (5.68)
  Week 12: number analyzed (Participants) | 282 | 291
  Week 12 | 13.3 (6.14) | 14.3 (6.32)
  Week 24: number analyzed (Participants) | 257 | 263
  Week 24 | 12.8 (6.93) | 14.2 (6.37)
  Week 36: number analyzed (Participants) | 249 | 253
  Week 36 | 12.8 (6.68) | 13.7 (6.85)

4. Secondary Outcome: Opioid Use
Description: Morphine milligram equivalent per day (MME/day). A lower MME is better as this indicates less prescription opioid drug use. Lowest score: 0; Highest score: N/A
Time Frame: Weeks 12, 24, and 36
Population: Not all participants reported opioid use, as this was not an inclusion criterion but rather a subset of the study population. This outcome was assessed only for those participants reporting opioid use at the time of enrollment.
Measure: Mean (Standard Deviation); unit: morphine milliequivalents
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 53 | 64
morphine milliequivalents
  Baseline | 45 (148) | 24 (36)
  Week 12: number analyzed (Participants) | 43 | 55
  Week 12 | 47 (163) | 32 (53)
  Week 24: number analyzed (Participants) | 43 | 41
  Week 24 | 48 (165) | 29 (44)
  Week 36: number analyzed (Participants) | 39 | 45
  Week 36 | 49 (173) | 27 (43)

5. Secondary Outcome: Number of Falls
Description: Number of fall events per arm.
Time Frame: Throughout the 36-week follow-up
Measure: Number; unit: number of falls
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
number of falls | 138 | 155

6. Secondary Outcome: Rate of Falls
Description: Event rate as calculated by number of falls/patient years
Time Frame: Though Week 36 follow-up
Measure: Number; unit: falls/patient year
Arm/Group | Pain Coping Skills Training (PCST) | Usual Care
Number analyzed (Participants) | 319 | 324
falls/patient year | 0.66 | 0.70

7. Secondary Outcome: Number of Hospitalizations
Description: Number of hospitalizations per arm.
Time Frame: Through 36-week follow-up
Measure: Number; unit: hospitalizations
Arm/Group | Pain Coping Skills Training (PCST) | Usual Care
Number analyzed (Participants) | 319 | 324
hospitalizations | 349 | 313

8. Secondary Outcome: Rate of Hospitalizations
Description: Event rate as calculated by number of hospitalizations/patient years
Time Frame: Through Week 36 follow-up
Measure: Number; unit: hospitalizations/patient year
Arm/Group | Pain Coping Skills Training (PCST) | Usual Care
Number analyzed (Participants) | 319 | 324
hospitalizations/patient year | 1.67 | 1.42

9. Secondary Outcome: Number of Deaths
Description: The number of deaths per arms.
Time Frame: Through the 36-week follow-up
Measure: Number; unit: deaths
Arm/Group | Pain Coping Skills Training (PCST) | Usual Care
Number analyzed (Participants) | 319 | 324
deaths | 35 | 34

10. Secondary Outcome: Rate of Deaths
Description: Rate of deaths as calculated by number of events/patient years
Time Frame: Through Week 36 follow-up
Measure: Number; unit: deaths/patient year
Arm/Group | Pain Coping Skills Training (PCST) | Usual Care
Number analyzed (Participants) | 319 | 324
deaths/patient year | 0.17 | 0.15

11. Secondary Outcome: Buprenorphine Acceptability
Description: The proportion of participants who initiate buprenorphine from among those offered buprenorphine.
Time Frame: Through Week 36
Measure: Number; unit: proportion of participants
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
proportion of participants | .27 | .50

12. Secondary Outcome: Buprenorphine Tolerability
Description: The proportion of patients who started buprenorphine and did not discontinue buprenorphine due to adverse effects or intolerance.
Time Frame: Through Week 36
Measure: Number; unit: proportion of participants
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
proportion of participants | 1.00 | .33

13. Secondary Outcome: Overall Sense of Quality of Life
Description: Quality of life will be measured using the Single-Item Quality of Life (QOL) Scale (SIS) from McGill Quality of Life (MQOL) questionnaire. Lowest score - 0; highest score - 10; Higher score equals better outcome.
Time Frame: Weeks 12, 24, and 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
score on a scale
  Baseline | 6.08 (2.61) | 5.82 (2.68)
  Week 12: number analyzed (Participants) | 282 | 291
  Week 12 | 6.66 (2.53) | 5.88 (2.54)
  Week 24: number analyzed (Participants) | 256 | 263
  Week 24 | 6.70 (2.43) | 6.09 (2.46)
  Week 36: number analyzed (Participants) | 249 | 252
  Week 36 | 6.27 (2.70) | 6.19 (2.52)

14. Secondary Outcome: Physical Functioning
Description: Physical functioning will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Functioning Short Form (SF)-6b questionnaire. Normalized score reported as t-values. The full range of possible scores is 21-59. 50 indicates the population mean with a standard deviation of 10. A higher score represents a better outcome.
Time Frame: Weeks 12, 24, and 36
Population: Participants withdrew at various points during the study, and some participants were unable to complete the PRO assessments.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
T-score
  Baseline: number analyzed (Participants) | 318 | 323
  Baseline | 33.5 (7.60) | 33.3 (7.68)
  Week 12: number analyzed (Participants) | 278 | 287
  Week 12 | 35.5 (8.08) | 33.9 (7.59)
  Week 24: number analyzed (Participants) | 256 | 255
  Week 24 | 35.0 (8.40) | 34.2 (8.09)
  Week 36: number analyzed (Participants) | 239 | 250
  Week 36 | 34.9 (7.89) | 34.5 (8.47)

15. Secondary Outcome: Depression
Description: Depression will be measured using the Patient Health Questionnaire (PHQ)-9. Lowest score - 0; Highest score - 27; Lower score equals better outcome.
Time Frame: Weeks 12, 24, and 36
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
score on a scale
  Baseline: number analyzed (Participants) | 310 | 319
  Baseline | 8.78 (5.77) | 9.51 (6.11)
  Week 12: number analyzed (Participants) | 277 | 278
  Week 12 | 7.29 (5.22) | 8.92 (5.83)
  Week 24: number analyzed (Participants) | 255 | 255
  Week 24 | 7.47 (5.90) | 8.96 (5.72)
  Week 36: number analyzed (Participants) | 245 | 245
  Week 36 | 8.29 (6.04) | 8.75 (6.09)

16. Secondary Outcome: Anxiety
Description: Anxiety will be measured using the Generalized Anxiety Disorder (GAD)-7 questionnaire. Lowest score - 0; Highest score - 21; Lower score equals better outcome.
Time Frame: Weeks 12, 24, and 36
Population: Participants withdrew at various points throughout the trial, and some participants were unable to complete the PRO assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
score on a scale
  Baseline: number analyzed (Participants) | 319 | 321
  Baseline | 6.76 (5.84) | 7.38 (6.14)
  Week 12: number analyzed (Participants) | 281 | 288
  Week 12 | 5.63 (5.48) | 7.04 (6.03)
  Week 24: number analyzed (Participants) | 257 | 259
  Week 24 | 6.18 (5.83) | 7.48 (5.89)
  Week 36: number analyzed (Participants) | 245 | 253
  Week 36 | 6.22 (5.75) | 6.96 (6.09)

17. Secondary Outcome: Coping
Description: Coping will be measured using the 1-Item Coping Strategies Questionnaire (CSQ). Lowest score - 0; Highest score - 6; Lower score equals better outcome.
Time Frame: Weeks 12, 24, and 36
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
score on a scale
  Baseline | 3.19 (2.19) | 3.50 (2.29)
  Week 12: number analyzed (Participants) | 282 | 291
  Week 12 | 2.56 (2.07) | 2.90 (2.11)
  Week 24: number analyzed (Participants) | 258 | 259
  Week 24 | 2.50 (2.16) | 2.86 (2.11)
  Week 36: number analyzed (Participants) | 246 | 252
  Week 36 | 2.41 (2.15) | 2.62 (2.06)

18. Secondary Outcome: Sleep Quality
Description: Sleep quality will be measure using the PROMIS Sleep Disturbance Short Form (SF) 6a.
  Normalized score reported as t-values. The full range of possible scores is 31.7 - 76.1. 50 indicates the population mean with a standard deviation of 10. A lower score represents a better outcome.
Time Frame: Weeks 12, 24, and 36
Population: Participants withdrew at various times during the study, and some participants were unable to complete the PRO assessments.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
t-score
  Baseline: number analyzed (Participants) | 314 | 322
  Baseline | 57.3 (9.95) | 58.2 (10.3)
  Week 12: number analyzed (Participants) | 276 | 285
  Week 12 | 54.3 (11.5) | 57.4 (9.94)
  Week 24: number analyzed (Participants) | 253 | 258
  Week 24 | 54.2 (10.9) | 56.8 (10.3)
  Week 36: number analyzed (Participants) | 243 | 252
  Week 36 | 54.3 (11.2) | 55.9 (11.1)

19. Secondary Outcome: Fatigue
Description: Fatigue will be measured using the PROMIS Fatigue Short Form (SF) 6a. Normalized score reported as t-values. The full range of possible scores is 26.2 - 65.6. 50 indicates the population mean with a standard deviation of 10. A lower score represents a better outcome.
Time Frame: Weeks 12, 24, and 36
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
t-score
  Baseline: number analyzed (Participants) | 317 | 319
  Baseline | 59.0 (10.0) | 59.4 (9.82)
  Week 12: number analyzed (Participants) | 274 | 286
  Week 12 | 56.2 (11.4) | 58.4 (10.7)
  Week 24: number analyzed (Participants) | 253 | 255
  Week 24 | 56.6 (12.0) | 58.4 (10.7)
  Week 36: number analyzed (Participants) | 242 | 247
  Week 36 | 57.0 (11.1) | 57.5 (10.8)

20. Secondary Outcome: Satisfaction With Treatment
Description: Satisfaction will be measured using the Patient Global Impression of Change (PGIC). Lowest score - 1; Highest score - 7; Lower score equals better outcome.
Time Frame: Weeks 12, 24, and 36
Population: Participants withdrew at various times throughout the trial, and some participants were unable to complete the PRO assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
score on a scale
  Week 12: number analyzed (Participants) | 281 | 289
  Week 12 | 3.10 (1.28) | 4.02 (1.37)
  Week 24: number analyzed (Participants) | 257 | 259
  Week 24 | 3.16 (1.42) | 3.69 (1.36)
  Week 36: number analyzed (Participants) | 245 | 251
  Week 36 | 3.16 (1.38) | 3.63 (1.47)

21. Secondary Outcome: Social Support
Description: Social support will be measured using the Multidimensional Scale of Perceived Social Support (MSPSS). Lowest score - 1; Highest score - 7; Higher score is better and equals more support. Total score reported.
Time Frame: Weeks 12, 24, and 36
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
score on a scale
  Baseline: number analyzed (Participants) | 311 | 322
  Baseline | 5.29 (1.46) | 5.02 (1.54)
  Week 12: number analyzed (Participants) | 267 | 282
  Week 12 | 5.37 (1.41) | 5.18 (1.42)
  Week 24: number analyzed (Participants) | 249 | 250
  Week 24 | 5.43 (1.33) | 5.26 (1.28)
  Week 36: number analyzed (Participants) | 237 | 243
  Week 36 | 5.38 (1.35) | 5.20 (1.39)

22. Secondary Outcome: Family Intrusion
Description: Family intrusion will be measured using the PROMIS Satisfaction with Social Roles and Activities. Normalized score reported as t-values. The full range of possible scores is 26.2 - 65.6. 50 indicates the population mean with a standard deviation of 10. A higher score represents a better outcome.
Time Frame: Weeks 12, 24, and 36
Population: Participants withdrew at various times during the study. Some participants were unable to complete the PRO assessments.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
T-score
  Baseline: number analyzed (Participants) | 318 | 319
  Baseline | 42.8 (9.29) | 43.3 (9.57)
  Week 12: number analyzed (Participants) | 277 | 288
  Week 12 | 44.4 (9.71) | 43.8 (9.22)
  Week 24: number analyzed (Participants) | 252 | 257
  Week 24 | 45.1 (9.67) | 43.9 (9.27)
  Week 36: number analyzed (Participants) | 244 | 248
  Week 36 | 44.5 (10.3) | 42.9 (9.77)

23. Secondary Outcome: Self-Efficacy
Description: Self-efficacy will be measured using the PROMIS Self-Efficacy for Managing Chronic Conditions - Managing Symptoms - Short Form 8A and the Single item targeting self-efficacy for pain.
  PROMIS Self-Efficacy for Managing Chronic Conditions - Managing Symptoms - Short Form 8A: Lowest score - 8; Highest score - 40; Higher score equals better outcome.
  Normalized score reported.
  Single item targeting self-efficacy for pain: Lowest score - 0; Highest score - 100; Higher score equals better outcome.
Time Frame: Weeks 12, 24, and 36
Population: Participants withdrew at various times during the study. Some participants were unable to complete the PRO assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
score on a scale
  Baseline: number analyzed (Participants) | 318 | 317
  Baseline | 45.4 (8.11) | 45.1 (8.32)
  Week 12: number analyzed (Participants) | 281 | 288
  Week 12 | 48.1 (8.75) | 46.2 (7.55)
  Week 24: number analyzed (Participants) | 256 | 258
  Week 24 | 48.3 (9.17) | 46.6 (8.79)
  Week 36: number analyzed (Participants) | 245 | 251
  Week 36 | 48.1 (9.10) | 47.2 (8.75)

24. Secondary Outcome: Presence of Other Symptoms
Description: Presence of symptoms will be measured using the Dialysis Symptom Index (DSI) Symptom Subscale. Lowest score - 0; Highest score - 30; Lower score equals better outcome.
Time Frame: Weeks 12, 24, and 36
Population: Participants withdrew at various points during the study. Not all participants were able to complete the PRO assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
score on a scale
  Baseline: number analyzed (Participants) | 314 | 315
  Baseline | 15.8 (6.39) | 16.5 (6.45)
  Week 12: number analyzed (Participants) | 276 | 285
  Week 12 | 14.3 (6.80) | 15.8 (6.38)
  Week 24: number analyzed (Participants) | 250 | 251
  Week 24 | 14.2 (6.80) | 15.8 (6.68)
  Week 36: number analyzed (Participants) | 243 | 243
  Week 36 | 14.3 (7.03) | 15.0 (7.01)

25. Secondary Outcome: Severity of Other Symptoms
Description: Severity of symptoms will be measured using the Dialysis Symptom Index (DSI) Symptom Subscale. Lowest score - 0; Highest score - 150; Lower score equals better outcome.
Time Frame: Week 12, 24, 36
Population: Participants withdrew at various times during the trial. Not all participants were able to complete the PRO assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
score on a scale
  Baseline: number analyzed (Participants) | 310 | 312
  Baseline | 55.2 (27.5) | 58.2 (27.3)
  Week 12: number analyzed (Participants) | 270 | 283
  Week 12 | 48.4 (28.3) | 55.9 (28.7)
  Week 24: number analyzed (Participants) | 247 | 247
  Week 24 | 48.9 (28.9) | 54.8 (28.0)
  Week 36: number analyzed (Participants) | 240 | 241
  Week 36 | 48.7 (28.0) | 51.9 (29.1)

26. Secondary Outcome: Discrimination
Description: Discrimination will be measured using the Everyday Discrimination Scale Short Version (EDS-S). Lowest score - 0; Highest score - 5; Lower score equals better outcome.
Time Frame: Baseline, Week 36
Population: Participants withdrew at various times during the study. Some participants were unable to complete the PRO assessments.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pain Coping Skills Training | Usual Care
Number analyzed (Participants) | 319 | 324
score on a scale
  Baseline: number analyzed (Participants) | 315 | 323
  Baseline | 4.75 (4.70) | 4.76 (4.95)
  Week 36: number analyzed (Participants) | 244 | 245
  Week 36 | 3.86 (4.70) | 4.18 (5.23)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of 36 Weeks, beginning after consent.
Arm/Group | Pain Coping Skills Training | Usual Care
All-Cause Mortality (participants affected / at risk) | 35/319 | 34/324
Serious Adverse Events (participants affected / at risk) | 169/319 | 167/324
Other Adverse Events (participants affected / at risk) | 102/319 | 115/324
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pain Coping Skills Training (N=319) | Usual Care (N=324)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 8 (9)
Cardiac arrest (Cardiac disorders) | 7 (8) | 7 (8)
Volume overload (Metabolism and nutrition disorders) | 24 (28) | 21 (25)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 7 (7)
COVD-19 (Infections and infestations) | 8 (8) | 19 (20)
Pneumonia (Infections and infestations) | 18 (20) | 6 (7)
Fall (Injury, poisoning and procedural complications) | 17 (19) | 26 (27)
AV graft complication (Injury, poisoning and procedural complications) | 0 (0) | 7 (10)
Kidney transplant (Surgical and medical procedures) | 8 (8) | 5 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 12 (16) | 22 (27)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (6) | 6 (6)
Gastroparesis (Gastrointestinal disorders) | 2 (6) | 1 (4)
Stroke (Nervous system disorders) | 8 (8) | 5 (6)
Suicidal ideation (Psychiatric disorders) | 2 (7) | 1 (2)
Hypertension (Vascular disorders) | 17 (21) | 13 (17)
Hypotension (Vascular disorders) | 12 (15) | 10 (10)
choledocolithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Peritoneal carcinomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (9)
abdominal pain (Gastrointestinal disorders) | 4 (4) | 3 (3)
acute mesenteric ischemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
acute toxic metabolic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
altered mental status (Psychiatric disorders) | 1 (1) | 0 (0)
ambulatory dysfunction (General disorders) | 2 (2) | 0 (0)
amputation (Surgical and medical procedures) | 6 (7) | 4 (4)
angina (Cardiac disorders) | 1 (1) | 1 (1)
angioplasty (Surgical and medical procedures) | 3 (3) | 2 (2)
anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
ascites (Gastrointestinal disorders) | 0 (0) | 1 (2)
assault (Social circumstances) | 1 (1) | 0 (0)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
atherosclerosis (Vascular disorders) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 5 (5) | 5 (6)
AV heart block (Cardiac disorders) | 1 (1) | 0 (0)
AV fistula complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
AV fistula placement (Surgical and medical procedures) | 0 (0) | 2 (2)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
bacteremia (Infections and infestations) | 10 (14) | 8 (9)
bed bugs (Social circumstances) | 1 (1) | 0 (0)
bladder infection (Infections and infestations) | 1 (1) | 0 (0)
blod clot (Vascular disorders) | 0 (0) | 3 (3)
blood infection (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
bowel obstruction (Gastrointestinal disorders) | 2 (2) | 3 (3)
bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
brain infarct (Nervous system disorders) | 0 (0) | 1 (1)
bronchial inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
c. diff (Infections and infestations) | 4 (6) | 2 (2)
CABG (Surgical and medical procedures) | 2 (2) | 0 (0)
car accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
cardiac ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
cardiac catheterization (Investigations) | 3 (3) | 2 (2)
cellulitis (Infections and infestations) | 2 (2) | 7 (8)
chest pain (Musculoskeletal and connective tissue disorders) | 10 (15) | 5 (5)
cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
coronary artery disease (Cardiac disorders) | 2 (2) | 1 (2)
critical limb ischemia (Vascular disorders) | 2 (2) | 0 (0)
diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
decreased cardiac function (Cardiac disorders) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
dental abscess (Infections and infestations) | 0 (0) | 1 (1)
diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (7) | 0 (0)
diabetic necrotizing infection (Infections and infestations) | 0 (0) | 1 (1)
diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
dialysis (Surgical and medical procedures) | 0 (0) | 1 (1)
dialysis access complication (Injury, poisoning and procedural complications) | 25 (32) | 15 (18)
dialysis access creation (Surgical and medical procedures) | 3 (3) | 1 (1)
dialysis access infection (Infections and infestations) | 8 (8) | 0 (0)
dialysis access revision (Surgical and medical procedures) | 1 (3) | 1 (1)
dialysis access surgery (Surgical and medical procedures) | 0 (0) | 1 (2)
diverticulitis (Infections and infestations) | 3 (5) | 1 (1)
dizziness (Nervous system disorders) | 2 (2) | 0 (0)
duodenal avm (Vascular disorders) | 0 (0) | 1 (1)
duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
DVT (Vascular disorders) | 1 (2) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 7 (7)
e. coli (Infections and infestations) | 1 (1) | 0 (0)
elevated INR (Investigations) | 0 (0) | 1 (1)
encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
endocarditis (Infections and infestations) | 2 (2) | 1 (1)
enlarged pulmonary artery (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
enlarged scrotum (Reproductive system and breast disorders) | 1 (1) | 0 (0)
enterococcus (Infections and infestations) | 1 (1) | 0 (0)
ESRD (Renal and urinary disorders) | 2 (2) | 0 (0)
eye surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
femoral bypass surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
fever (General disorders) | 2 (2) | 0 (0)
fistulogram (Investigations) | 0 (0) | 1 (1)
flu (Infections and infestations) | 2 (2) | 1 (1)
folliculitis (Infections and infestations) | 0 (0) | 1 (1)
foot infection and pain (Infections and infestations) | 3 (6) | 2 (2)
fracture (Injury, poisoning and procedural complications) | 12 (12) | 6 (6)
gallbladder infection (Infections and infestations) | 1 (1) | 0 (0)
gangrene (Infections and infestations) | 0 (0) | 3 (3)
gastrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastric ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
GI bleed (Gastrointestinal disorders) | 4 (4) | 5 (5)
Grave's Disease (Immune system disorders) | 1 (1) | 0 (0)
h. pylori infection (Infections and infestations) | 1 (1) | 0 (0)
hand injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
hand pain and infection (Infections and infestations) | 3 (3) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 0 (0)
hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
heart attack (Cardiac disorders) | 3 (3) | 3 (3)
heart blockage (Cardiac disorders) | 0 (0) | 1 (1)
heart failure (Cardiac disorders) | 3 (3) | 8 (8)
heart surgery (Surgical and medical procedures) | 1 (1) | 4 (4)
heart valve replacement (Surgical and medical procedures) | 3 (3) | 0 (0)
hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
hemorrhagic shock (Vascular disorders) | 1 (1) | 0 (0)
hemorrhoids (Gastrointestinal disorders) | 1 (2) | 1 (1)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hernia (General disorders) | 0 (0) | 1 (1)
hernia repair (Surgical and medical procedures) | 2 (2) | 0 (0)
hidradenitis axillaris (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hidradenitis suppurativa (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HIV (Infections and infestations) | 0 (0) | 1 (1)
hospitalization (Surgical and medical procedures) | 0 (0) | 1 (1)
hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypervolemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypervolemic hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypovolemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
ICA stenosis (Nervous system disorders) | 0 (0) | 1 (1)
ileostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
urine retention (Renal and urinary disorders) | 0 (0) | 1 (2)
infection (Infections and infestations) | 4 (4) | 6 (6)
inguinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
INR instability (Investigations) | 0 (0) | 1 (1)
internal defibrillator complication (Product Issues) | 0 (0) | 1 (1)
intraventricular hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
ischemic colitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
IVC clot (Vascular disorders) | 1 (1) | 0 (0)
ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
kidney infection (Infections and infestations) | 0 (0) | 2 (2)
kidney failure (Renal and urinary disorders) | 0 (0) | 2 (2)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
liver disease (Hepatobiliary disorders) | 1 (1) | 1 (1)
liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
lower extremity swelling (General disorders) | 1 (1) | 0 (0)
mania (Psychiatric disorders) | 1 (1) | 0 (0)
mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
mesenteric thrombophlebitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
metabolic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
metabolic instability (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
metapneumovirus (Infections and infestations) | 1 (1) | 0 (0)
MRSA (Infections and infestations) | 1 (1) | 0 (0)
myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
necrosis (General disorders) | 0 (0) | 1 (1)
nephrectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
neutrophic keratitis (Eye disorders) | 0 (0) | 1 (1)
non-traumatic L hyphema (Eye disorders) | 0 (0) | 1 (1)
NSTEMI (Cardiac disorders) | 6 (6) | 2 (2)
osteomyelitis (Infections and infestations) | 3 (4) | 7 (7)
pain (General disorders) | 0 (0) | 1 (1)
pancreatitis (Gastrointestinal disorders) | 2 (7) | 2 (3)
paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
parathyroidectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
pemphigus foliaceus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4)
percutaneous intervention (Surgical and medical procedures) | 1 (1) | 0 (0)
pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1)
pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
peripheral artery disease (Vascular disorders) | 0 (0) | 3 (3)
peripheral neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
peritonitis (Infections and infestations) | 1 (1) | 0 (0)
pinched nerve (Nervous system disorders) | 1 (1) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (4)
pneumonitis (Infections and infestations) | 0 (0) | 1 (1)
polycystic disease (Renal and urinary disorders) | 0 (0) | 1 (1)
polypharmacy (Investigations) | 1 (1) | 0 (0)
prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
pseudogout (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
pubic ramus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
seizure (Nervous system disorders) | 1 (1) | 0 (0)
sepsis (Infections and infestations) | 8 (8) | 3 (3)
septic shock (Infections and infestations) | 0 (0) | 3 (3)
shingles (Infections and infestations) | 0 (0) | 1 (1)
shock (Vascular disorders) | 3 (3) | 0 (0)
shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
sickle cell disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
sigmoid ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (9)
somnolence (Nervous system disorders) | 1 (1) | 0 (0)
spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
stab wounds (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
staph infection (Infections and infestations) | 1 (1) | 1 (1)
Steal Syndrome (Vascular disorders) | 0 (0) | 1 (1)
STEMI (Cardiac disorders) | 1 (1) | 1 (1)
streptococcus (Infections and infestations) | 1 (1) | 0 (0)
subgaleal hematoma (Vascular disorders) | 1 (1) | 0 (0)
subdural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
surgery (Surgical and medical procedures) | 10 (10) | 6 (6)
syncope (Nervous system disorders) | 1 (1) | 2 (2)
tachycardia (Cardiac disorders) | 1 (1) | 5 (5)
tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
thrombectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
ulcerative lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
unconsciousness (Nervous system disorders) | 2 (2) | 0 (0)
upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
urinary tract infection (Infections and infestations) | 1 (1) | 6 (7)
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
volume shifts (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 8 (10) | 1 (1)
weakness (General disorders) | 0 (0) | 3 (3)
wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pain Coping Skills Training (N=319) | Usual Care (N=324)
Withdrawal symptoms (General disorders) | 1 | 5
Suicidal ideation (Psychiatric disorders) | 11 | 19
Adverse effect from a medication starting to treat pain, depression or anxiety (General disorders) | 11 | 9
Fall (Injury, poisoning and procedural complications) | 84 | 94
Opioid use disorder (Psychiatric disorders) | 0 | 0
Substance use disorder (Psychiatric disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT04571619/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT04571619/ICF_002.pdf